CLINICAL TRIAL: NCT00479635
Title: A Phase II Trial of TPI 287 in Patients With Metastatic Prostate Cancer Who Have Progressive Neoplastic Disease Following Treatment With One Prior Taxane Regimen
Brief Title: A Phase II Trial of TPI 287 in Patients With Metastatic Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor could no longer support; enrollment stopped August 2008.
Sponsor: Cortice Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPI 287-04
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Prostate Cancer
Keywords: HRPC; TPI 287; Taxane; MDR; Hormone Refractory Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — TPI-287

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TPI 287 (Experimental)
  Interventions: Drug: TPI 287

INTERVENTIONS:
Drug: TPI 287 — 160 mg/m2 every three weeks for six cycles
Drug: TPI 287 — 160 mg/m2 intravenously over 60 minutes every three weeks until toxicity or progression of disease.

SUMMARY:
The primary objective of the study is to determine the response rate to TPI 287 in patients with metastatic, hormone-refractory prostate cancer who have had one prior taxane regimen.

DETAILED DESCRIPTION:
This is an open-label, multi-center, 2-stage Simon design, Phase 2 study of TPI 287 in patients with metastatic, hormone-refractory prostate cancer. All patients must have received prior taxane therapy. Up to 80 patients will be enrolled and stratified based on duration of cumulative exposure to a single prior taxane regimen. A single taxane regimen is considered to he a taxane or taxane containing therapy administered on a defined schedule with no more than 2 months' interruption between treatments, and total exposure will be assessed by the number of months on that schedule.

One stratum (up to 40 patients) will consist of patients who have had over 3 months (up to a maximum of 10 months) exposure to a taxane regimen, who then have documented progression of disease (initially taxane sensitive). The second stratum (up to 40 patients) will consist of patients considered primarily resistant to taxanes who have had documented progressive disease as best response after exposure to a single taxane regimen for less than or equal to 3 months. Patients may have received prior hormonal therapy and/or bisphosphonates and may continue on these therapies.

In the first stage of the trial, 22 patients in each stratum will be treated with TPI 287 intravenously every 21 days. If 1 or fewer patients in either stratum demonstrate a response in this first stage, the trial will be discontinued for that stratum. Otherwise, an additional 18 patients in the stratum showing 2 or more responses will be enrolled in the second stage of the study. If 4 or fewer patients demonstrate a response in the total study population in either stratum from stages 1 and 2, then the drug will not be considered of interest in prostate cancer for patients as defined in that stratum.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological evidence of adenocarcinoma of the prostate and have metastatic disease.
* Patients must have received only one prior regimen for their advanced disease. This regimen must have included a taxane.

  * First Stratum Eligibility: Patients must have advanced, metastatic prostate cancer with documented progression after receiving more than three months of treatment, up to a total of 10 months with 1 prior taxane regimen. Prior best response to treatment, and duration of response, will be recorded.
  * Second Stratum Eligibility: Patients must have advanced, metastatic prostate cancer that has progressed as best response despite three months or less of treatment with 1 prior taxane regimen.
* Must have castrate levels of testosterone less than 50 ng/mL
* Must have an ECOG Performance Score of 0 or 1
* Must be age 18 or older
* Must be able to read, understand and sign informed consent
* Serum creatinine less than or equal to 2.0 mg/dL
* Total bilirubin less than or equal to 2.0 mg/dL
* SGOT/SGPT less than or equal to 3 times the ULN
* ANC greater than or equal to 1500/UL
* Platelet count greater than or equal to 100,000/UL Recovered from the effects of prior surgery, radiotherapy or other antineoplastic therapy.

Exclusion Criteria:

* Active infection or with a fever greater than or equal to 38.5 degrees centigrade within 3 days of first scheduled day of dosing
* More than one prior systemic therapy for HRPC beyond androgen-ablative therapy. Prior systemic therapy may have been administered for metastatic disease or as adjuvant therapy
* Has received radiotherapy to greater than 30% of their active bone marrow
* History of prior malignancy within the past 5 years except for curatively treated non-melanoma skin cancer
* Impending fracture of a weight bearing bone
* Known hypersensitivity to any of the components of TPI 287
* Receiving concurrent investigational therapy or who have received investigational therapy within 30 days of study start
* Grade 2 peripheral neuropathy
* NYHA Class 3 or 4 congestive heart failure
* Any medial condition that would interfere with ability to sign ICF, cooperate and participate in the study or interfere with interpretation of results
* History of allogenic transplant
* Know HIV or Hepatitis B or C positive

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Response | 15 months

SECONDARY OUTCOMES:
Time to progression | 15 months
Duration of response | 6 months
Safety | Continuous

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Silberman, MD, PhD, Study Director — SLS Oncology, LLC
Locations (6):
- United States (6):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Comprehensive Cancer Center at Desert Mountain, Palm Springs, California
  - University of Kentucky, Lexington, Kentucky
  - Kansas City Cancer Center South, Kansas City, Missouri
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- See also: Related Info — http://www.archerbio.com/